CLINICAL TRIAL: NCT03899077
Title: A Phase II Study Comparing Salvage Radiotherapy in Combination With 6 Months of Androgen-deprivation Therapy Versus Anti-androgen Therapy With Apalutamide in Patients With Biochemical Progression After Radical Prostatectomy
Brief Title: Radiotherapy Combined With a LHRH (Ant)Agonist Versus Apalutamide in Patients With Biochemical Recurrence After RP
Acronym: SAVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research Antwerp (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTOR18001GZA
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Leuprolide; Powders; Goserelin; Injections, Subcutaneous; Triptorelin Pamoate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): The standard hormonal treatment in combination with salvage radiotherapy is ADT by a LHRH agonist or antagonist for 24 weeks. LHRH agonists and antagonists include leuprolide, goserelin, triptorelin, and degarelix.
  Interventions: Drug: Leuprorelin Acetate 45Mg Powder for Injection Suspension Vial; Drug: Goserelin Acetate 10.8 MG Subcutaneous Implant; Drug: Triptorelin Pamoate; Drug: Degarelix acetate
- Arm B (Experimental): Patients will receive 6 cycles (each cycle is 30 days) of the study drug (4x 60mg tablets daily in a single intake).
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — Apalutamide 240mg daily for 6 months (i.e. 6 28-day cycles); oral use
  Arms: Arm B
Drug: Leuprorelin Acetate 45Mg Powder for Injection Suspension Vial — Leuprorelin acetate 45mg for 6 months; subcutaneous use
  Arms: Arm A
Drug: Goserelin Acetate 10.8 MG Subcutaneous Implant — Goserelin acetate 10.8mg for 6 months; subcutaneous use
  Arms: Arm A
Drug: Triptorelin Pamoate — Triptorelin pamoate 22.5mg for 6 months; intramuscular use
  Arms: Arm A
Drug: Degarelix acetate — Degarelix acetate 80mg for 6 months; subcutaneous use
  Arms: Arm A

SUMMARY:
This is a phase II randomized, open-label study comparing salvage radiotherapy in combination with 6 months of androgen-deprivation therapy (ADT) with LHRH agonist or antagonist (arm A) versus anti-androgen therapy (AAT) with apalutamide 240mg daily (arm B) in hormone-naïve patients with biochemical progression after radical prostatectomy. All subjects will receive salvage radiotherapy as standard of care and will be randomly assigned in a 1:1 ratio to receive either 6 months of androgen-deprivation therapy (ADT) with LHRH agonist or antagonist through 6 monthly, two 3-monthly or one 6-monthly injections (control arm) or 6 28-day cycles of apalutamide 240mg daily (interventional arm). The study will include a screening phase, treatment phase, and a post-treatment phase. The primary objective of the trial is to compare sexual function between the 2 groups based on the Expanded Prostate cancer Index Composite (EPIC)-26 sexual domain scores at 9 months after start of hormonal treatment.

DETAILED DESCRIPTION:
After radical prostatectomy, around one third of patients will have biochemical progression. Salvage radiotherapy (SRT) is still potentially curative, but about 40-50% of patients will progress further. Recently, success rates of SRT were significantly improved through the use of concomitant anti-androgen (AAT) or androgen-deprivation (ADT) therapy. In RTOG 96-01, 2 years of bicalutamide 150 mg resulted in a 5% overall survival benefit at 12-years. In GETUG-AFU 16, 5-year progression-free survival was significantly improved when SRT was combined with 6 months of an LHRH agonist. Based on GETUG-AFU 16, most radiation oncologists now combine SRT with at least 6 months of ADT. However, ADT comes with several serious side-effects, both physical (cardiovascular, metabolic, musculoskeletal) and psychological (sexual, emotional and cognitive). It appears worthwile to look for alternatives in the form of AAT. In that respect, apalutamide, a potent competitive and purely antagonistic second-generation anti-androgen, is the ideal candidate.

This trial is a phase II randomized, open-label study comparing salvage radiotherapy in combination with 6 months of ADT (arm A) versus AAT with apalutamide 240mg daily (arm B) in hormone-naïve patients with biochemical progression after radical prostatectomy. All subjects will receive salvage radiotherapy as standard of care and will be randomly assigned in a 1:1 ratio to receive either 6 months of ADT with LHRH agonist or antagonist through 6 monthly, two 3-monthly or one 6-monthly injections (control arm A) or 6 28-day cycles of apalutamide 240mg daily (interventional arm B).

The study will include a screening phase, treatment phase, and a post-treatment phase.

1. Screening phase: allows for assessment of subject eligibility up to 35 days prior to randomization.
2. Treatment phase: includes the hormonal treatment for 6 months, to be started at the most 2 weeks after randomization and standard salvage radiotherapy. During the treatment phase, patients will have 3 study visits:

   1. treatment initiation visit: first injection of LHRH (ant)agonist (arm A) or cycle 1, day 1 (C1D1) of apalutamide (arm B).
   2. Concurrent with RT visit: if necessary (depending on product prescribed) injection of LHRH (ant)agonist (arm A) or cycle 4, day 1 (C4D1) of apalutamide (arm B).
   3. End of treatment visit: at the end of the 6 months of hormonal therapy.
3. Post-treatment phase: will begin after a subject completes the treatment phase and the end of treatment visit and will continue until the primary endpoint is reached, i.e. the 9-months (3 months after end of treatment visit) EPIC-26 sexual domain score.

The primary objective of the trial is to compare sexual function between the 2 groups based on the EPIC-26 sexual domain (0 - 100 scale, with higher scores representing better sexual function) at 9 months after start of hormonal treatment (primary endpoint). The following secondary endpoints will be explored:

1. Quality of life: assessed using EPIC-26 as well as the EORTC quality of life questionnaires C30 and PR25 as well as FACT-P.
2. Toxicity: will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
3. Efficacy: prostate-specific antigen (PSA) response rates, defined as a decline from baseline in PSA level of 80% or greater, as well as PSA complete response rates, defined as a decline from baseline in PSA level of 90% or greater, will be prospectively collected at the 4 treatment visits.

At this point in time, no study has directly compared apalutamide to LHRH agonists or antagonists in combination with SRT. This trial may be a preamble to the design of a registration trial in such patients or indeed patients with a intermediate and high-risk localized disease that are scheduled for EBRT or brachytherapy as radical treatment and also benefit from 6 months of hormonal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male, > 18 years old.
2. ECOG 0-1.
3. Histologically confirmed adenocarcinoma of the prostate.
4. Previous radical prostatectomy (RP), pT2-3, pN0 or pNx.
5. PSA detectable with confirmed rise (at least 2 weeks apart) at least 8 weeks after RP.
6. Hormone-naive disease.
7. Patients amendable to take oral medication.
8. Patients must have clinical laboratory values at screening:

   1. Hemoglobin 9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
   2. Platelet count ≥100,000 x 109/µL independent of transfusion and/or growth factors within 3 months prior to randomization
   3. Serum albumin ≥3.0 g/dL
   4. Serum creatinine <2.0 × upper limit of normal (ULN)
   5. Serum potassium ≥3.5 mmol/L
   6. Serum total bilirubin 1.5 × ULN (note: in subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, subject may be eligible)
   7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5 × ULN
9. Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry.
10. Patient agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
11. Patients who have received the information sheet and signed the informed consent form.
12. Patients must be willing to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with severe erectile dysfunction according to international index of erectile function (IIEF-5) questionnaire (score 1-7).
2. Allergies, hypersensitivity or known intolerance to the study drugs or excipients.
3. History of any of the following:

   1. Seizure or known condition that may pre-dispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to randomization, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect).
   2. Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization.
4. Current evidence of any of the following:

   1. Uncontrolled hypertension.
   2. Gastrointestinal disorder affecting absorption.
5. Patients already included in another clinical trial involving an experimental drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
EPIC-26 sexual domain score | 9 months after start of hormonal treatment
  EPIC-26 sexual domain score (0 - 100 scale, with higher scores representing better sexual function)

SECONDARY OUTCOMES:
FACT-P quality of life global score | 9 months after start of hormonal treatment
  Health related quality of life (QoL) will be assessed using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire designed for patients with prostate cancer. It consists of 27 core items which assess patient function in four domains: physical, social/family, emotional, and functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain, as well as a global QoL score. Higher scores represent better QoL.
EORTC QLQ C30 quality of life score | 9 months after start of hormonal treatment
  Quality of life will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) C30. The EORTC QLQ-C30 contains 30 items and is composed of both multi-item scales and single- item measures. These include five functional scales (physical, role, emotional, cognitive and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/QoL scale.
EORTC QLQ PR25 quality of life score | 9 months after start of hormonal treatment
  Quality of life will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) PR25. scale. The EORTC QLQ-PR25 is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 25 items specifically related to prostate cancer.
Grade of acute toxicity | After obtaining informed consent and up to 30 days after last dose
  Acute as well as late toxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (published November 27, 2017)
PSA response rates | 0, 3, 6, and 9 months
  Prostate-specific antigen (PSA) response rates, defined as a decline from baseline in PSA level of 80% or greater, as well as PSA complete response rates, defined as a decline from baseline in PSA level of 90% or greater, will be prospectively collected at 0, 3, 6, and 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Piet Dirix, Principal Investigator — Gasthuis Zusters Antwerpen
Locations (9):
- Belgium (9):
  - OLVZ Aalst, Aalst
  - AZ Sint-Jan, Bruges
  - Hopital Erasme, Brussels
  - UZ Gent, Ghent
  - CH Jolimont, Haine-Saint-Paul
  - UZ Brussel, Jette
  - AZ Groeninge, Kortrijk
  - CHU UCL Namur, Namur
  - GZA, Wilrijk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dirix P, Strijbos M, den Mooter TV, Liefhooghe N, Bruwaene SV, Uvin P, Ghysel C, Ost D, Schatteman P, Bral S, Engels B, den Begin RV, Otte FX, Roumeguere T, Palumbo S, Neybuch Y, Fonteyne V, Ost P, Dirix L. Phase II open-label study investigating apalutamide in patients with biochemical progression after radical prostatectomy. Future Oncol. 2020 Jun;16(16):1083-1189. doi: 10.2217/fon-2020-0056. Epub 2020 May 1. PMID 32356465